CLINICAL TRIAL: NCT05866523
Title: Teamwork Makes the Dream Work: Team-based Inpatient Anti-Retroviral Treatment and Access to Services (ARTAS)
Brief Title: Teamwork Makes the Dream Work
Acronym: ARTAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 5230236
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Inpatient Facility Diagnoses
Keywords: HIV, linkage to care, hospital readmission
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a prospective, observational cohort study design with patients enrolled at Loma Linda University Medical Center (LLUMC), evaluating a multidisciplinary inpatient linkage to care program compared to historical control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Historic Control (Active Comparator): Control group will get treatment as usual, which consists of medical care by primary admitting service
  Interventions: Behavioral: Standard of Care
- Team based inpatient ARTAS (Active Comparator): Eligible patients after the study consent process will receive Antiretroviral Treatment Access Study (ARTAS) intervention by social-worker and a medical consultation by an infectious disease physician
  Interventions: Behavioral: Team Based Inpatient ARTAS

INTERVENTIONS:
Behavioral: Team Based Inpatient ARTAS — Infectious Disease Team will provide inpatient consultation. Social Work Team will provide 1 session of case management inpatient and up to 5 case management sessions within 90 days post discharge or until the client is linked to medical care as evidenced by visit with HIV specialist within 90 days post discharge.
  Arms: Team based inpatient ARTAS
Behavioral: Standard of Care — Subject admitted and seen by routine inpatient medical service.
  Arms: Standard of Care Historic Control

SUMMARY:
Exploring the effect of team-based ARTAS intervention in an inpatient setting on HIV linkage to care and hospital readmission rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* newly diagnosed HIV
* Known diagnosis of HIV not on ART within 30 days of admission
* Known HIV and not virally suppressed based on interview
* Known HIV and has not been under the care of an HIV specialist within the past 6 months

Exclusion Criteria:

* All three criteria must be present for exclusion:
* virally suppressed
* actively taking ART
* are under active care of an HIV specialist within the last 6 months
* Less than 18 years of age (stand alone exclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of linkage to HIV care post discharge | Up to 90 days post-study enrollment hospitalization discharge
  Subject had one visit with HIV specialist post hospital discharge. This will be determined per medical chart review and phone interview with subject

SECONDARY OUTCOMES:
Readmission Rate after initial post-study hospitalization | Up to 90 days post-study enrollment hospitalization discharge
  Subject had one emergency room visit or one inpatient admission post hospital discharge. This will be determined per medical chart review and phone interview with subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craw JA, Gardner LI, Marks G, Rapp RC, Bosshart J, Duffus WA, Rossman A, Coughlin SL, Gruber D, Safford LA, Overton J, Schmitt K. Brief strengths-based case management promotes entry into HIV medical care: results of the antiretroviral treatment access study-II. J Acquir Immune Defic Syndr. 2008 Apr 15;47(5):597-606. doi: 10.1097/QAI.0b013e3181684c51. PMID 18285714
- [Background] Gardner LI, Metsch LR, Anderson-Mahoney P, Loughlin AM, del Rio C, Strathdee S, Sansom SL, Siegal HA, Greenberg AE, Holmberg SD; Antiretroviral Treatment and Access Study Study Group. Efficacy of a brief case management intervention to link recently diagnosed HIV-infected persons to care. AIDS. 2005 Mar 4;19(4):423-31. doi: 10.1097/01.aids.0000161772.51900.eb. PMID 15750396
- [Background] Gardner LI, Marks G, Craw J, Metsch L, Strathdee S, Anderson-Mahoney P, del Rio C; Antiretroviral Treatment Access Study Group. Demographic, psychological, and behavioral modifiers of the Antiretroviral Treatment Access Study (ARTAS) intervention. AIDS Patient Care STDS. 2009 Sep;23(9):735-42. doi: 10.1089/apc.2008.0262. PMID 19645619